CLINICAL TRIAL: NCT04624425
Title: Additional Effects of Segmental Breathing In Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00710 Asma Baig
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Asthma; Segmental Breathing
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmental breathing exercises (Experimental): Segmental breathing exercises, Treatment session will be last for 10-15 minutes. For 2 Weeks
  Interventions: Other: Segmental breathing exercises
- Buteyko breathing exercises (Active Comparator): Buteyko breathing exercises, Treatment session will be last for 10-15 minutes. For 2 Weeks
  Interventions: Other: Buteyko breathing exercises

INTERVENTIONS:
Other: Segmental breathing exercises — Segmental breathing exercises along with the Conventional Treatment of buteyko breathing exercises for two weeks of duration. Segmental breathing exercises include 18-20 breaths in one session (6 breaths/min) with rest interval after every 6 breaths.
  Arms: Segmental breathing exercises
Other: Buteyko breathing exercises — Buteyko exercises for two weeks of duration. Treatment session will be last for 10-15minutes.
  Arms: Buteyko breathing exercises

SUMMARY:
To determine the effects of segmental breathing exercise and buteyko breathing exercises on chest expansion in individuals with asthma. To determine the effects of segmental breathing exercise and buteyko breathing exercises on pulmonary function (FEV1, FVC, FEV1/FVC) in individuals with asthma. To determine the effects of segmental breathing exercise and buteyko breathing exercises on Asthma Control Questionnaire in individuals with asthma.

DETAILED DESCRIPTION:
The National Heart and Lung Institute determines asthma as a common chronic airway disease distinguished by variable and reoccurring manifestations, bronchial hypersensitivity, reducing the flow of air in and out of the lungs and inflammatory reactions with in air passages in the lungs.

Earlier in the first place asthma is also defined as existence of spontaneously reversible airway obstruction or with treatment and narrowing of airways also increased to different stimuli i.e. abrupt changes in weather, cold air, histamine, dust, pollen, feathers, exercise, viral upper respiratory infection, animal dander, cigarette smoke, fungal spores or respiratory allergens that increases bronchial hypersensitivity.

segmental breathing technique is used for increasing the expansion of chest in individual's having empyema whose expansion has been decreased. Total 40 individuals with empyema were included in this study. Chest expansion at three levels have been checked i.e. at axilla level, at sternum level and at xiphoid level were examined before and after implementation of segmental exercise technique. Segmental breathing techniques play a major role in expansion of damaged lungs and as a consequence integral to rehabilitation of Respiratory disease.

The effectiveness of segmental breathing technique and deep breathing exercise on expansion of chest and pulmonary function test. The physical therapy treatment comprises of dyspnea alleviating positions, simple breathing exercises, and exercises for thoracic expansion, inspiratory muscle training with incentive spirometers. Segmental breathing techniques are used to give support or enhance expansion of restricted lung in respiratory disorder. This technique is meant to have an effect on variation of mechanism, involving the stretch reflex process. Fast stretch on external intercostal muscles brings on assistance in contraction.

Intercostal stretching with breathing control exercises might be more effective in enhancing lung parameters. This may also take part in ventilator capacity like tidal volume, saturation of oxygen and minute ventilation. Intercostal stretching might have stimulated the receptors of stretch mechanism in chest wall, hence distend the thoracic cavity which would have connected to medulla oblongata with nerve cell.

The efficacy of buteyko method on control of asthma and quality of living in individuals with asthma. The buteyko breathing exercise is non-medical method that had shown to be better in reducing the frequency and seriousness of asthma. The interventional group manifested a considerable improvement in control of asthma score and quality of living score after four weeks. The other control group didn't manifest any improvement. This study suggested that buteyko breathing exercise may upgrade the physical, societal, spiritual and occupational effect on asthma and improved quality of living.

The combined effect of buteyko breathing exercise and walking exercise on peak expiratory flow. The experimental group was specified for the combination of buteyko exercises and walking exercise for duration of eight weeks, three times per week and of 55 minutes of training session. The benefit of this technique is hold interval that can decrease overuse of carbon dioxide (CO2) that will control breath rate with the help of medulla oblongata in respiratory center, providing Nitric oxide (NO) which particular has bronchodilator effect. These both exercises minimise inflammatory reaction so that they decrease the sign and symptoms of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical diagnosis of asthma.

Exclusion Criteria:

* Participants with unbearable chest pain, chylothorax, hemothorax, pneumothorax.
* Participants with pleura disorder and chest trauma & rib fracture.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 2 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 2 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Modified Borg Scale of Perceived Exertion | 2 weeks
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.
Chest Expansion measurement at Axillary level | 2 weeks
  A measuring tape with centimeters scale will be used for measuring the expansion at Axillary level. Changes from the baseline will be measured.
Chest Expansion measurement at Spinal cord T4 level | 2 weeks
  A measuring tape with centimeters scale will be used for measuring the expansion at at Spinal cord T4 level. Changes from the baseline will be measured.
Chest Expansion measurement at xiphoid process | 2 weeks
  A measuring tape with centimeters scale will be used for measuring the expansion at xiphoid process level. Changes from the baseline will be measured.
Asthma Control Questionnaire | 2 weeks
  Measurement of the adequateness of asthma control and modifications in asthma control which may occurs immediately or as a consequence of treatment. It is a 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%). Scores range between 0 (totally controlled) and 6 (severely uncontrolled) .The 7-items Asthma Control Questionnaire (ACQ) is valid to measure the goals of asthma management as defined by international guideline. Changes from the baseline will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Nusrat Abdul Rauf Centre for Enablement (NACE), Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No